CLINICAL TRIAL: NCT05228834
Title: A Phase 3b, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Treatment Effect of Voxelotor on Neurocognitive Function in Pediatric Participants 8 to < 18 Years of Age With Sickle Cell Disease
Brief Title: Voxelotor Neurocognitive Function Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Data will not inform further development of Voxelotor
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBT440-044; C5341028 (Other: Alias Study Number)
Record Dates: First submitted 2022-01-10; First posted 2022-02-08 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-03

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Drug (Experimental): Voxelotor 1500mg or equivalent daily as a tablet or powder for oral suspension
  Interventions: Drug: Voxelotor Only Product in Oral Dose Form
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Voxelotor Only Product in Oral Dose Form — During the Randomized Treatment Period, participants will be randomized in a 1:1 ratio to receive 1500 mg of voxelotor (or the weight-adjusted equivalent dose for participants < 12 years old), once daily (administered orally as tablets/PFOS) or matching placebo for 12 weeks in addition to ongoing standard of care (SOC) treatment.
  Arms: Active Drug
Drug: Placebo — During the Randomized Treatment Period, participants will be randomized in a 1:1 ratio to receive 1500 mg of voxelotor (or the weight-adjusted equivalent dose for participants < 12 years old), once daily (administered orally as tablets/PFOS) or matching placebo for 12 weeks in addition to ongoing standard of care (SOC) treatment.
  Arms: Placebo

SUMMARY:
This is a Phase 3b, randomized, double-blind, placebo-controlled, multicenter study to assess the treatment effect of voxelotor on neurocognitive function as assessed by the National Institute of Health (NIH) Toolbox Cognition Module of executive abilities in pediatric participants (8 to < 18 years) with SCD.

DETAILED DESCRIPTION:
Eligible participants will receive daily treatment with 1500 mg voxelotor or matching placebo for 12 weeks. During screening and at the end of 12 weeks participants will undergo a series of tests to measure the change in neurocognitive functions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants with confirmed diagnosis of SCD (all genotypes). Documentation of SCD genotype is required and may be based on documented history of laboratory testing or confirmed by laboratory testing during Screening.
2. Aged 8 to < 18 years.
3. Screening Hb level 5.5 to 10.5 g/dL.
4. Able to answer NIH Toolbox Module questions validated and normed based on age and maternal education on tablet.
5. If participant is receiving HU they must have been on a stable dose for at least 90 days prior to signing the ICF/AF, with no dose modifications or initiation of HU planned or anticipated by the Investigator.
6. If participant is receiving erythropoiesis-stimulating agents (ESAs) they must have been on a stable dose for at least 12 weeks before enrollment with no dose modifications planned or anticipated by the Investigator.
7. Participants, who if female and of child-bearing potential, agree to use highly effective methods of contraception from study start to 30 days after the last dose of study drug and who if male, agree to use barrier methods of contraception and refrain from donating sperm from study start to 30 days after the last dose of study drug.
8. Females of child-bearing potential must have a negative pregnancy test before the administration of study drug.
9. Parental/guardian consent and participant assent (between ≥ 12 and < 18 years) per Institutional Review Board (IRB)/Independent ethics committee (IEC) policy and requirements, consistent with International Council for Harmonisation (ICH) guidelines.
10. Capable of complying with the requirements and restrictions in the protocol, and willing to participate in the study.

Exclusion Criteria:

1. Receiving chronic transfusion therapy.
2. Red blood cell (RBC) transfusion within 3 months before initiation of study drug or receives scheduled RBC transfusion therapy (also termed chronic, prophylactic, or preventive transfusion).
3. History of overt stroke including hemorrhagic stroke or transient ischemic attack (TIA) or spinal cord injury, magnetic resonance angiography (MRA)-defined vasculopathy, or magnetic resonance imaging (MRI)/transcranial doppler (TCD)-documented silent cerebral infarcts.
4. Congenital brain malformation, previously diagnosed severe developmental disability (eg, autism and/or intelligence quotient [IQ] < 60, and/or severe attention deficit hyperactivity disorder [ADHD]), or impairment that would prevent the use of a computer tablet.
5. Participant is taking or has received voxelotor (Oxbryta®) within 90 days prior to the Screening Visit.
6. Surgery within 8 weeks before Day 1 or planned elective surgery during the study.
7. Anemia due to bone marrow failure (eg, myelodysplasia).
8. Absolute reticulocyte count (ARC) < 100 × 10^9/L.
9. Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 4× upper limit of normal (ULN).
10. Severe renal dysfunction (estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m^2) or is on chronic dialysis.
11. Clinically significant bacterial, fungal, parasitic, or viral infection which requires therapy.

    1. Patients with acute bacterial infection requiring antibiotic use should delay screening /enrollment until the course of antibiotic therapy has been completed.
    2. Patients with known active hepatitis A, B, or C or who are known to be human immunodeficiency virus (HIV) positive.
12. Symptomatic coronavirus disease of 2019 (COVID-19) infection.
13. Females who are breast-feeding or pregnant.
14. History of hematopoietic stem cell transplant or gene therapy.
15. Participants taking concomitant medications such as sensitive cytochrome P450 (CYP)3A4 substrates with a narrow therapeutic range, or strong CYP3A4 inducers
16. Participated in another clinical trial of an investigational product (or medical device) within 30 days or 5 half-lives of date of informed consent, whichever is longer, or is currently participating in another trial of an investigational product (or medical device).
17. Medical, psychological, or behavioral condition that, in the opinion of the Investigator, would confound or interfere with evaluation of safety and/or efficacy of the study drug, prevent compliance with the study protocol; preclude informed consent; or, render the participant unable/unlikely to comply with the study procedures.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-044

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 1 participant was enrolled. The study was terminated due to slow enrollment and resource reprioritization at Global Blood Therapeutics (L-GBT). Based on the low enrollment, data was not reported due to risk of re-identification of participant.
Groups:
- Voxelotor: Participants were to be randomized to receive Voxelotor 1500 milligram (mg) orally once daily for 12 weeks.
- Placebo: Participants were to be randomized to receive placebo matched to Voxelotor 1500 mg orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Voxelotor | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only one participant was enrolled. Hence, data cannot be reported due to risk of re-identification of participant.
Groups:
- Voxelotor: Participants were to be randomized to receive Voxelotor 1500 mg orally once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Voxelotor | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Customized [unit: Participants]
Sex: Female, Male [unit: Participants]
Race/Ethnicity, Customized [unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Executive Abilities Composite Score Assessed Using NIH Toolbox Cognition Module At Week 12
Description: The NIH toolbox cognition module is a standardized cognitive battery comprising of executive function, episodic memory, language, processing speed, working memory, and attention as subdomains. The toolbox is comprised of 7 test instruments that measure 8 abilities within 6 major cognitive domains and have been categorized as executive abilities (Dimensional Change Card Sort Test, Flanker Inhibitory Control and Attention Test, and List Sorting Test) and nonexecutive abilities (Picture Vocabulary Test, Oral Reading Recognition Test, and Picture Sequence Memory Test). The NIH toolbox standard score has a mean of 100 and standard deviation (SD) of 15. The higher the score, the better the performance.
Time Frame: Baseline (last assessment prior to first dose of study treatment), Week 12
Population: Study was terminated and only one participant was enrolled. Hence, data cannot be reported for this outcome measure due to risk of re-identification of participant.
Arm/Group | Voxelotor | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in Pattern Comparison Processing Speed Test Scores Assessed Using NIH Toolbox Cognition Module at Week 12
Description: The NIH Toolbox Cognition Battery Test is a comprehensive set of neuro behavioral measurements used to assess cognitive, sensory and motor functions where a higher composite score equals better cognitive performance. The NIH Toolbox Cognitive Scores used the Fully Adjusted Scale score (also referred to as the fully corrected T-score) with a mean of 50 and standard deviation of 10.
Time Frame: Baseline (last assessment prior to first dose of study treatment), Week 12
Population: as for outcome 1
Arm/Group | Voxelotor | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Nonexecutive Cognitive Abilities Composite Score Assessed Using NIH Toolbox Cognition Module Up to Week 12
Description: The NIH toolbox cognition module is a standardized cognitive battery comprising of executive function, episodic memory, language, processing speed, working memory, and attention as subdomains. The toolbox is currently comprised of 7 test instruments that measure 8 abilities within 6 major cognitive domains and have been categorized as executive abilities (Dimensional Change Card Sort Test, Flanker Inhibitory Control and Attention Test, and List Sorting Test) and nonexecutive abilities (Picture Vocabulary Test, Oral Reading Recognition Test, and Picture Sequence Memory Test). Baseline was defined as the last assessment performed prior to receiving the first dose of study treatment. The NIH toolbox standard score has a mean of 100 and SD of 15. The higher the score, the better the performance.
Time Frame: Baseline (last assessment prior to first dose of study treatment) up to Week 12
Population: as for outcome 1
Arm/Group | Voxelotor | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Hemoglobin Level Up to Week 12
Time Frame: Baseline (last assessment prior to first dose of study treatment) up to Week 12
Population: as for outcome 1
Arm/Group | Voxelotor | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count Up to Week 12
Time Frame: Baseline (last assessment prior to first dose of study treatment) up to Week 12
Population: as for outcome 1
Arm/Group | Voxelotor | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Percentage Reticulocyte Up to Week 12
Time Frame: Baseline (last assessment prior to first dose of study treatment) up to Week 12
Population: as for outcome 1
Arm/Group | Voxelotor | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase (LDH) Up to Week 12
Time Frame: Baseline (last assessment prior to first dose of study treatment) up to Week 12
Population: as for outcome 1
Arm/Group | Voxelotor | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Unconjugated Bilirubin Up to Week 12
Time Frame: Baseline (last assessment prior to first dose of study treatment) up to Week 12
Population: as for outcome 1
Arm/Group | Voxelotor | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percent Change From Baseline in Unconjugated Bilirubin, Absolute Reticulocyte, Percentage Reticulocytes, Lactate Dehydrogenase (LDH) Up to Week 12
Time Frame: Baseline (last assessment prior to first dose of study treatment) up to Week 12
Population: as for outcome 1
Arm/Group | Voxelotor | Placebo
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event was defined as any untoward medical occurrence associated with the use of a drug in participants whether or not considered drug related. TEAEs were those events with onset dates that occurred during the treatment period.
Time Frame: From start of study treatment (Day 1) up to Week 12
Population: as for outcome 1
Arm/Group | Voxelotor | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not reported.
Description: Study was terminated and only one participant was enrolled. Hence, data cannot be reported due to risk of re-identification of participant.
Arm/Group | Voxelotor | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated due to slow enrollment and resource reprioritization at L-GBT. Based on the low enrolment data was not reported due to risk of re-identification of participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT05228834/Prot_SAP_000.pdf